CLINICAL TRIAL: NCT01830088
Title: Family-based Treatment of Depressed Adolescents: An Empirical Study With Norwegian Adolescents in Specialty Mental Health Care
Brief Title: Family Based Treatment of Depressed Adolescents (AHUS)
Acronym: BudFam2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding period expired before reaching recruitment goal.
Sponsor: University Hospital, Akershus (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Helse Sor-Ost (Other Government); University of Oslo (Other)
Responsible Party: Principal Investigator, Marianne Villabo, Researcher, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BudFam2
Record Dates: First submitted 2013-04-08; First posted 2013-04-12 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Depressive Disorder; Mood Disorder; Major Depression
MeSH Terms: conditions — Depressive Disorder; Mood Disorders; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: The two treatment arms are i) Attachment Based Family Therapy and ii) Treatment as usual
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors (HAM-D) are masked and do not know the treatment arm of the participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attachment Based Family Therapy (Experimental): Attachment-Based Family Therapy (ABFT) is primarily a process oriented, emotion focused treatment guided by a semi-structured treatment protocol. ABFT aims to improve the family's capacity for problem solving, affect regulation, and organization. This strengthens family cohesion which can buffer against depression, suicidal thinking, and risk behaviors
  Interventions: Behavioral: Attachment Based Family Therapy
- Enhanced Usual Care (Active Comparator): No attempt is made to control any aspect of the enhanced usual care except for pre-scheduled assessment plan
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Attachment Based Family Therapy — Attachment-Based Family Therapy (ABFT) is is primarily a process oriented, emotion focused treatment guided by a semi-structured treatment protocol. ABFT aims to improve the family's capacity for problem solving, affect regulation, and organization. This strengthens family cohesion which can buffer against depression, suicidal thinking, and risk behaviors
  Other Names: ABFT
  Arms: Attachment Based Family Therapy
Behavioral: Enhanced Usual Care — No attempt is made to control any aspect of the enhanced usual care except for pre-scheduled assessment plan
  Other Names: EUC
  Arms: Enhanced Usual Care

SUMMARY:
Major depressive disorder (MDD) affects about 5% of adolescents and is on the rise both internationally and in Norway. Further, it is also associated with increased risk for suicide. Not surprisingly, depression is the largest reason for referral to specialty mental health services for adolescents (13-17 years) in Norway. Although anti-depressants and Cognitive behavioral therapy are strong treatments and have received extensive research, the best treatments show a recovery rate of only 37 %.

There is a need to develop and test alternative treatments that can stand alone or augment anti-depressant medication. Family factors play an important role in the etiology, maintenance and relapse of depression. A promising family-based treatment (Attachment based family therapy- ABFT) was imported to Norway and its feasibility tested in a pilot randomized clinical trial with 20 families. The results showed promising treatment outcomes. Although the developers of the model have refined, adapted the model to suicidal ideation and built strong technology to support dissemination, a definitive study of ABFT for adolescents with major depression has not yet been conducted. Therefore the primary aim of this study is to test if ABFT is more effective that enhanced usual care (EUC) to treat clinic-referred adolescents with major depression. The investigators will test the hypothesis that 12 weeks of ABFT therapy will produce a greater proportion of adolescents report remission from depression and symptom change than 12 weeks of enhanced clinical care (EUC). Secondary research aims are i) to test a hypothesis that parent-adolescent conflict will be more sensitive to change for adolescents receiving ABFT that adolescents receiving EUC ii) to explore patterns of change in suicidal ideation in the recruited sample in the acute-phase treatment.

Central challenges to the study are i) blinding therapists/patients, which is difficult in psychotherapy trials ii) lack of a standardized control condition, and iii) selecting and training regular staff therapists to high adherence levels. However, with tighter control over these factors than is normal for a typical effectiveness trial, the investigators expect results to show what to expect under the "best of conditions" in community clinics. Benchmark derived from the study will inform how to effectively train therapists and subsequently implement the model into mainstream services.

ELIGIBILITY:
Inclusion criteria:

* Adolescents between ages 13-17 years
* Adolescents endorsing depression symptoms (HAM-D ≥ 16) on the HAM-D
* Adolescents meet diagnostic criteria for major depressive disorder (MDD) as assessed by Kiddie SADS
* At least one primary parent or caregiver must participate in the assessment and treatment

Exclusion criteria:

* psychotic disorder
* anorexia nervosa
* severe substance dependence disorders
* mental retardation (IQ less than 70 as assessed by the clinician)
* asperger syndrome/autism as assessed by the K-SADS
* Adolescents taking antidepressant medication for depression for less than 6 weeks prior to the screening

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2013-10; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Hamilton Depression Rating scale | 12, 24 and 48 weeks
  The Hamilton Depression Rating Scale (17 item) version is a 17-item, semi-structured interview and is currently a widely used clinical measure depression. Grid HamD (Williams 2008) version is used.

SECONDARY OUTCOMES:
Beck depression Inventory (BDI-II) | Bi-weekly for 12 weeks, and at week 24 and week 48
Kiddie-SADS (Diagnostic interview) | Baseline and 26 weeks

OTHER OUTCOMES:
Change from baseline in Conflict Behavior Questionnaire | Biweekly for 12 weeks and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Marianne A Villabø, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lorenskog, Akershus, Norway

REFERENCES:
- [Background] Israel P, Diamond GS. Feasibility of Attachment Based Family Therapy for depressed clinic-referred Norwegian adolescents. Clin Child Psychol Psychiatry. 2013 Jul;18(3):334-50. doi: 10.1177/1359104512455811. Epub 2012 Aug 28. PMID 22930777
- [Derived] Waraan L, Rognli EW, Czajkowski NO, Aalberg M, Mehlum L. Effectiveness of attachment-based family therapy compared to treatment as usual for depressed adolescents in community mental health clinics. Child Adolesc Psychiatry Ment Health. 2021 Feb 12;15(1):8. doi: 10.1186/s13034-021-00361-x. PMID 33579332